CLINICAL TRIAL: NCT01506297
Title: Biologic Assessment of Satiety
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC504
Record Dates: First submitted 2012-01-03; First posted 2012-01-09 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: obesity; satiety; body weight management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Subjective measures of satiety are correlated with biologic mechanisms of appetite control.

ELIGIBILITY:
Inclusion Criteria:

* medical history (interview) demonstrating good health
* non-smoking
* not taking steroid-based medications
* not planning to or currently attempting to gain or lose weight
* being willing to consent to study conditions
* healthy adults ages 25-45 years
* body mass index between 18-30 kg/m2.
* University of North Dakota students may participate but student status is not required.

Exclusion Criteria:

* diagnosed eating disorders
* current or planned pregnancy
* lactation
* unmanaged hypertension (systolic >160 mmHg or diastolic > 100mmHg) and/or other cardiovascular, pulmonary, skeletal and metabolic diseases
* taking medications known to affect appetite, body composition, weight, or food intake

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Correlation of subjective and objective satiety responses | measures at -30, -15, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240, 300 minutes
  Comparison of subjective responses and gut hormone responses of satiety

SECONDARY OUTCOMES:
Repeatability of subjective and objective measures of satiety | measures at -30, -15, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240, 300 minutes
  Repeated assessment (3 times) of subjective and objective responses to food intake

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Raatz, PhD, Principal Investigator — USDA GFHNRC
Locations (1):
- USDA Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No